CLINICAL TRIAL: NCT02442271
Title: An Open-Label, Multicenter Study to Evaluate the Efficacy and Safety of Ombitasvir/ABT-450/Ritonavir and Dasabuvir With or Without Ribavirin (RBV) in Treatment-Naïve or Treatment-Experienced Adults in Brazil With Genotype 1 Chronic Hepatitis C Virus (HCV) Infection (TOPAZ III)
Brief Title: A Study to Evaluate the Efficacy and Safety of Three Experimental Drugs in Adults With Hepatitis C Virus Infection, Who Are Either Treatment-naive or Treatment-experienced in Brazil
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-225
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Results first posted 2017-08-01 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Chronic Hepatitis C Infection
Keywords: Chronic Hepatitis C; Hepatitis C Treatment Naive; Hepatitis C Genotype 1; Hepatitis C Treatment Experienced; Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — ombitasvir; dasabuvir; Viekira Pak; paritaprevir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 3-DAA ± RBV (Experimental): 3-DAA (ombitasvir/paritaprevir/ritonavir [25 mg/150 mg/100 mg once daily] and dasabuvir [250 mg twice daily]) with or without weight-based ribavirin (± RBV; dosed 1,000 or 1,200 mg daily divided twice a day) for 12 or 24 weeks.
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir and dasabuvir; Drug: ribavirin

INTERVENTIONS:
Drug: ombitasvir/paritaprevir/ritonavir and dasabuvir — Tablet; ombitasvir coformulated with paritaprevir and ritonavir, dasabuvir tablet
  Other Names: Viekira Pak; paritaprevir also known as ABT-450; ombitasvir also known as ABT-267; dasabuvir also known as ABT-333
Drug: ribavirin — Tablet

SUMMARY:
The purpose of this study is to evaluate the proportion of subjects achieving sustained virologic response 12 weeks post-treatment (SVR12) in adults with genotype 1 (GT1) chronic HCV infection, who received treatment with 3 direct-acting antiviral agents (3-DAAs; ombitasvir/paritaprevir/ritonavir and dasabuvir) with or without ribavirin.

ELIGIBILITY:
Inclusion Criteria:

* Females must be post-menopausal for more than 2 years or surgically sterile or practicing acceptable forms of birth control
* Males must be surgically sterile or agree to practice acceptable forms of birth control
* Chronic hepatitis C virus (HCV) infection at screening
* Fibrosis stage F3 or greater, documented by acceptable tests
* Participants with cirrhosis: Absence of hepatocellular carcinoma (HCC) as indicated by acceptable methods

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Positive test result for Hepatitis B surface antigen (HbsAg) or anti-HIV antibody positive (HIV Ab)
* Use of contraindicated medications within 2 weeks of dosing
* Clinically significant abnormalities or co-morbidities
* History of solid organ transplant
* Abnormal laboratory tests
* Current or past clinical evidence of Child-Pugh B or C classification or clinical history of liver decompensation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2015-04-27 (Actual); Primary Completion 2016-07-04 (Actual); Study Completion 2016-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc, Study Director — AbbVie

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Treatment regimen was assigned according to HCV genotype/subtype and cirrhosis status.
Groups:
- 3-DAA ± RBV: 3-DAA (ombitasvir/paritaprevir/ritonavir [25 mg/150 mg/100 once daily] and dasabuvir [250 mg twice daily]) with or without weight-based ribavirin (± RBV; dosed 1,000 or 1,200 mg daily divided twice a day) for 12 or 24 weeks.
Period: Overall Study
Arm/Group | 3-DAA ± RBV
Started | 222
Completed | 218
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Withdrew Consent | 1
Not completed — Lost to Follow-up | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | 3-DAA ± RBV
Number analyzed (Participants) | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (10.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99
  Male | 123

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 12 weeks after the last dose of study drug. Participants with missing data were counted as failures.
Time Frame: 12 weeks after the last actual dose of study drug
Population: Intent-to-treat population: all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3-DAA ± RBV
Number analyzed (Participants) | 222
percentage of participants | 96.4 [93.1 to 98.2]

2. Secondary Outcome: Percentage of Participants With SVR12 by Fibrosis Stage
Description: SVR12 was defined as plasma HCV RNA level <LLOQ]12 weeks after the last dose of study drug. The percentage of participants achieving SVR12 by fibrosis stage (F3 and F4) are presented. Participants with missing data were counted as failures.
Time Frame: 12 weeks after the last actual dose of study drug
Population: All participants in the ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Fibrosis Stage F3: Participants with baseline fibrosis stage F3 (without cirrhosis).
- Fibrosis Stage F4: Participants with baseline fibrosis stage F4 (with compensated cirrhosis).
Arm/Group | Fibrosis Stage F3 | Fibrosis Stage F4
Number analyzed (Participants) | 89 | 133
percentage of participants | 96.6 [90.6 to 98.8] | 96.2 [91.5 to 98.4]

3. Secondary Outcome: Percentage of Participants With SVR12 by Participant Prior HCV Treatment Experience
Description: SVR12 was defined as HCV RNA level <LLOQ 12 weeks after the last dose of study drug. Data are presented by prior HCV treatment experience. Data are provided by participants' prior HCV treatment experience at screening. Participants with missing data were counted as failures.
Time Frame: 12 weeks after the last actual dose of study drug
Population: All participants in the ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Treatment-Naive: Participants who had never received any antiviral treatment for HCV infection.
- Pegylated Interferon (PegIFN)/RBV Null Responders; Pegylated Interferon (PegIFN)/RBV Non-Responders: Participants who had received prior treatment with pegIFN-based therapy for HCV infection and failed to achieve a 1 log10 IU/mL reduction in HCV RNA by Week 4 or a 2 log10 IU/mL reduction in HCV RNA by Week 12 during a prior IFN/RBV or pegIFN/RBV treatment course
- Pegylated Interferon (PegIFN)//RBV Partial Responders: Participants who had received prior treatment with pegIFN-based therapy for HCV infection and achieved at least a 2 log10 IU/mL reduction in HCV RNA by Week 12 during a prior IFN/RBV or pegIFN/RBV treatment course but failed to achieve HCV RNA undetectable at the end of treatment
- Pegylated Interferon (PegIFN)/RBV Relapser: Participants who had received prior treatment with pegIFN-based therapy for HCV infection who achieved HCV undetectable at end of a prior IFN/RBV or pegIFN/RBV treatment course but HCV RNA was detectable following cessation of therapy
- Pegylated Interferon (PegIFN)/RBV Breakthrough: Participants who had received prior treatment with pegIFN-based therapy for HCV infection and achieved at least one documented result of HCV RNA undetectable during a prior IFN/RBV or pegIFN/RBV treatment course
- IFN Interolerant: Participants who did not meet any of the other definitions of treatment failure and discontinued IFN/RBV or pegIFN/RBV therapy due to IFN intolerability
- Other: Participants who received IFN treatment, including IFN or pegIFN monotherapy, IFN/RBV, or pegIFN/RBV experienced subjects. Includes subjects who do not have adequate documentation of response.
Arm/Group | Treatment-Naive | Pegylated Interferon (PegIFN)/RBV Null Responders | Pegylated Interferon (PegIFN)//RBV Partial Responders | Pegylated Interferon (PegIFN)/RBV Non-Responders | Pegylated Interferon (PegIFN)/RBV Relapser | Pegylated Interferon (PegIFN)/RBV Breakthrough | IFN Interolerant | Other
Number analyzed (Participants) | 102 | 22 | 7 | 26 | 34 | 12 | 7 | 12
percentage of participants | 96.1 [90.3 to 98.5] | 95.5 [78.2 to 99.2] | 100 [NA to NA] — The number of participants analyzed is <10 | 100 [87.1 to 100.0] | 97.1 [85.1 to 99.5] | 100 [78.5 to 100.00] | 85.7 [NA to NA] — The number of participants analyzed is <10 | 91.7 [64.6 to 98.5]

4. Secondary Outcome: Percentage of Participants With SVR12 by Participant Eligibility for Treatment With Interferon (IFN) at Screening
Description: SVR12 was defined as HCV RNA level <LLOQ 12 weeks after the last dose of study drug. Data are presented by prior HCV treatment experience. Data are provided by participants' eligibility for treatment with IFN at screening. Participants with missing data were counted as failures.
Time Frame: 12 weeks after the last actual dose of study drug
Population: All participants in the ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Interferon (IFN)-Ineligible, Treatment-Naive: Participants who had never received any antiviral treatment for HCV infection and were ineligible for treatment with IFN at screening.
- Interferon (IFN)-Eligible, Treatment-Naive: Participants who had never received any antiviral treatment for HCV infection and were eligible for treatment with IFN at screening.
- Interferon (IFN)-Ineligible, Treatment-Experienced: Participants who had received prior antiviral treatment for HCV infection and were ineligible for treatment with IFN at screening.
- Interferon (IFN)-Eligible, Treatment-Experienced: Participants who had received prior antiviral treatment for HCV infection and were eligible for treatment with IFN at screening.
Arm/Group | Interferon (IFN)-Ineligible, Treatment-Naive | Interferon (IFN)-Eligible, Treatment-Naive | Interferon (IFN)-Ineligible, Treatment-Experienced | Interferon (IFN)-Eligible, Treatment-Experienced
Number analyzed (Participants) | 10 | 92 | 7 | 113
percentage of participants | 90.0 [59.6 to 98.2] | 96.7 [90.8 to 98.9] | 85.7 [NA to NA] — The number of participants analyzed is <10 | 97.3 [92.5 to 99.1]

5. Secondary Outcome: Hepatitis C Virus Patient-Reported Outcomes Instrument (HCV-PRO) Total Score: Change From Baseline to 12 Weeks After the Last Dose of Study Drug
Description: The HCV-PRO has been developed to capture the function and well-being impact of HCV conditions and treatment and contains 16 items important to HCV-infected patients; items were totaled to a summary score. Scores range from 0 to 100. A higher HCV-PRO score indicates a better state of health and a decrease from baseline represents worsening. If a participant answered at least 12 of the 16 items, the missing items were imputed with the mean score of the answered items; if a participant did not answer at least 12 of the items, the total score was considered missing.
Time Frame: Day 1 (Baseline), 12 weeks after the last actual dose of the study drug
Population: All participants in the ITT population with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fibrosis Stage F3 | Fibrosis Stage F4
Number analyzed (Participants) | 88 | 130
units on a scale
  SVR12 Not Achieved: number analyzed (Participants) | 3 | 4
  SVR12 Not Achieved | 0.5 (10.97) | 0.8 (10.64)
  SVR12 Achieved: number analyzed (Participants) | 85 | 126
  SVR12 Achieved | 3.8 (13.25) | 4.2 (15.72)

6. Secondary Outcome: Short-Form 36 Version 2 Health Survey (SF-36v2) Physical Component Summary (PCS) Scores: Change From Baseline to 12 Weeks After the Last Dose of Study Drug
Description: The SF-36v2 is a non-disease specific Health Related Quality of Life (HRQoL) instrument. The SF-36v2 comprises 36 total items (questions) targeting a subject's functional health and well-being in 8 domains (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health) with a recall period of four weeks. Domain scores are aggregated into a Physical Component Summary (PCS) score and a Mental Component Summary (MCS) score. SF-36v2 scores range from 1-100: higher scores indicate a better state of health and a decrease from baseline represents worsening. If a participant answered at least 50% of the items in a multi-item scale of the SF-36v2, the missing items were imputed with the average score of the answered items in the same domain. In cases where the participant did not answer at least 50% of the items, the score for that domain was considered missing. The SF-36v2 MCS and PCS scores were not computed if any domain
Time Frame: Day 1 (Baseline), 12 weeks after the last actual dose of the study drug
Population: All participants in the ITT population with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fibrosis Stage F3 | Fibrosis Stage F4
Number analyzed (Participants) | 87 | 131
units on a scale
  SVR12 Not Achieved: number analyzed (Participants) | 3 | 4
  SVR12 Not Achieved | -0.5 (9.22) | 1.3 (8.59)
  SVR12 Achieved: number analyzed (Participants) | 84 | 127
  SVR12 Achieved | 0.1 (6.42) | 2.1 (7.60)

7. Secondary Outcome: (SF-36v2) Mental Component Summary (MCS) Scores: Change From Baseline to 12 Weeks After the Last Dose of Study Drug
Description: The SF-36v2 is a non-disease specific Health Related Quality of Life (HRQoL) instrument. The SF-36v2 comprises 36 total items (questions) targeting a subject's functional health and well-being in 8 domains (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health) with a recall period of four weeks. Domain scores are aggregated into a PCS score and a MCS score. Scores SF-36v2 scores range from 1-100: higher scores indicate a better state of health and a decrease from baseline represents worsening. If a participant answered at least 50% of the items in a multi-item scale of the SF-36v2, the missing items were imputed with the average score of the answered items in the same domain. In cases where the participant did not answer at least 50% of the items, the score for that domain was considered missing. The SF-36v2 MCS and PCS scores were not computed if any domain was missing.
Time Frame: Day 1 (Baseline), 12 weeks after the last actual dose of the study drug
Population: All participants in the ITT population with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fibrosis Stage F3 | Fibrosis Stage F4
Number analyzed (Participants) | 87 | 131
units on a scale
  SVR12 Not Achieved: number analyzed (Participants) | 3 | 4
  SVR12 Not Achieved | 2.4 (3.72) | -0.6 (8.47)
  SVR12 Achieved: number analyzed (Participants) | 84 | 127
  SVR12 Achieved | 2.4 (11.39) | 2.5 (9.15)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until 30 days after the last dose of study drug (up to 28 weeks).
Description: TEAEs and TESAEs are defined as any AE or SAE with onset or worsening after the first dose of study drug until 30 days after the last dose of study drug.
Arm/Group | 3-DAA ± RBV
Serious Adverse Events (participants affected / at risk) | 6/222
Other Adverse Events (participants affected / at risk) | 139/222
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 3-DAA ± RBV (N=222)
DIARRHOEA (Gastrointestinal disorders) | 1
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 1
HEPATIC FAILURE (Hepatobiliary disorders) | 1
GASTROENTERITIS (Infections and infestations) | 1
LUNG ADENOCARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1
RENAL FAILURE (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 3-DAA ± RBV (N=222)
ANAEMIA (Blood and lymphatic system disorders) | 16
DIARRHOEA (Gastrointestinal disorders) | 19
DYSPEPSIA (Gastrointestinal disorders) | 15
NAUSEA (Gastrointestinal disorders) | 34
ASTHENIA (General disorders) | 20
FATIGUE (General disorders) | 41
HEADACHE (Nervous system disorders) | 48
INSOMNIA (Psychiatric disorders) | 12
COUGH (Respiratory, thoracic and mediastinal disorders) | 14
PRURITUS (Skin and subcutaneous tissue disorders) | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.